CLINICAL TRIAL: NCT02747173
Title: Study to Assess Bone Biomarkers for TKI Response in RCC Patients With Bone Metastasis and HRQoL in These Patients as Well as Comparing Whole Body MRI vs. Bone Scintigraphy and vs. CT in the Assessment of Metastatic Lesions
Brief Title: Assessment of Bone Biomarkers for TKI Response in RCC With Bone Metastases, HRQoL and Comparison of Imaging Techniques
Acronym: METHEOS
Status: Terminated | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: SOG-ANG-2014-01
Record Dates: First submitted 2015-04-23; First posted 2016-04-21 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Renal Cell Carcinoma
Keywords: metastatic, bone metastases
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RCC patients with bone metastases: Patients will receive the standard TKI treatment for first line treatment naive metastatic RCC. Sunitinib or pazopanib as decided by the investigator.

SUMMARY:
Prospective observational study to assess bone predictive biomarkers for TKI response in RCC patients with bone metastasis and HRQoL with TKI in these patients as well as the sensitivity and specificity of whole body magnetic resonance versus bone scintigraphy and versus CT in the assessment of metastatic lesions at bone level and at other sites.

DETAILED DESCRIPTION:
Prospective observational study to assess:

* Bone predictive biomarkers for tyrosine kinase inhibitor (TKI) response in renal cell carcinoma (RCC) patients with bone metastasis - Health Related Quality of Life (HRQoL) with TKI
* Comparison of the sensitivity and specificity of whole body magnetic resonance versus bone scintigraphy and versus Computerized tomography (CT) in the assessment of metastatic lesions at bone level and at other sites.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a stage IV renal cell carcinoma with confirmed presence of bone metastases, subsidiary of treatment with an TKI in first line
* 18 years old or more
* Life expectancy > 12 weeks
* Eastern Cooperative Oncology Group Performance Status (ECOG PS): 0 - 2
* Capability of understanding the study and completing the numerical pain scale, diary of analgesics and Quality of Life forms
* Patient who has given informed consent
* Adequate renal, hepatic and hematologic functions

Exclusion Criteria:

* Pregnancy, breastfeeding or fertile patients who do not use adequate contraceptive methods
* Non-clear cell histology
* Non irradiated brains metastases
* Symptomatic brain metastases
* Inability to undergo any of the medical tests of the study
* A history of breast cancer or melanoma. Other tumors are accepted as long as the patients has been for at least 5 years free of disease
* Synchronic diagnosis of another neoplasm
* Presence of an active infection
* Any decompensated disease or metabolic disorder
* Cardiac events or pulmonary embolism in the 12 months previous to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of a stage IV renal cell carcinoma with confirmed presence of bone metastases, subsidiary of treatment with an TKI in first line
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Assess bone biomarkers in response to TKI | Every 3 months until an average of 12 months
  Assess the predictive value to TKI of bone biomarkers (bone formation BAP, P1NP, OPG and osteocalcin, and bone resorption biomarkers CTX) in patients with RCC with bone metastases.

SECONDARY OUTCOMES:
Progression free survival | An average of 12 months
  Assess the efficacy of TKI in patients with RCC with bone metastases.
Objective response rate | An average of 12 months
  Assess the efficacy of TKI in patients with RCC with bone metastases.
Measurements in time of bone metastases in RCC using whole body magnetic resonance and bone scintigraphy | Every 3 months until an average of 12 months
  Comparison of the sensibility and specificity of whole body magnetic resonance and bone scintigraphy in the detection of metastases and response assessment of bone metastases in RCC
Change and correlation of magnetic resonance and CT results in the assessment of global disease response to TKI. Using RECIST and MASS criteria | Every 3 months until an average of 12 months
  Compare globally the magnetic resonance and CT results in the assessment of disease response to TKI using RECIST and MASS criteria
Quality of life of patients with RCC and bone metastases throughout the study period using the FSI-15 | Every 3 months until an average of 12 months
  Assess the quality of life of patients with RCC and bone metastases using the 15 item Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI-15)
Quality of life of patients with RCC and bone metastases throughout the study period using FACT-BP | Every 3 months until an average of 12 months
  Assess the quality of life of patients with RCC and bone metastases using the FACT-BP questionnaire
Efficacy of TKI in the improvement of pain produced by bone metastases throughout the study period | every week until an average of 12 months
  Assess the efficacy of TKI in the improvement of pain produced by bone metastases assessing the use of analgesics.
Efficacy of TKI in the improvement of pain produced by bone metastases throughout the study period using the NPR scale | every week until an average of 12 months
  Assess the efficacy of TKI in the improvement of pain produced by bone metastases using the Numeric Pain Rating Scale
Assessment osteonecrosis of the jaw with use of biphosphonates or denosumab throughout the study period | every week until an average of 12 months
  Risk of osteonecrosis of the jaw with use of biphosphonates or denosumab

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Vazquez, MD, Principal Investigator — Hospital Univ Lucus Augusti
Locations (12):
- Spain (12):
  - Hospital de Donostia, San Sebastián, Guipuzcoa
  - Complejo Hospitalario Univ de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Univ de Vigo, Vigo, Pontevedra
  - Hospital Universitario central de Asturias, Oviedo, Principality of Asturias
  - Consorcio Hospitalario Parc Tauli, Barcelona
  - Complejo Hospitalario de León, León
  - Hospital Univ Lucus Augusti, Lugo
  - Complejo Hospitalario de Ourense, Ourense
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza